CLINICAL TRIAL: NCT00906373
Title: A Multicenter, Phase 2 Study Evaluating IMC-A12 in Combination With Sorafenib as First-Line Therapy for Patients With Advanced Hepatocellular Carcinoma (HCC)
Brief Title: A Study of IMC-A12 in Combination With Sorafenib in Participants With Advanced Cancer of the Liver
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13931; CP13-0812 (Other: ImClone, LLC); I5A-IE-JAEG (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Results first posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Liver Neoplasms; Antibodies, Monoclonal
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — cixutumumab; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1, IMC A12 - 10 mg/kg (Active Comparator): Treatment cycles will repeat until there is evidence of progressive disease (PD), toxicity, or withdrawal. If any participant experiences a dose-limiting toxicity (DLT), an additional 3 participants will be enrolled at this dose level (for a total of 6). If no further DLTs, enrollment into Cohort 2 will occur.
  Interventions: Biological: IMC-A12 (cixutumumab) - 10 milligrams/kilogram (mg/kg); Drug: Sorafenib
- Cohort 2, IMC A12 20 - mg/kg (Active Comparator): Treatment cycles will repeat until there is evidence of PD, toxicity, or withdrawal.
  Interventions: Biological: IMC-A12 (cixutumumab) - 20 mg/kg; Drug: Sorafenib

INTERVENTIONS:
Biological: IMC-A12 (cixutumumab) - 10 milligrams/kilogram (mg/kg) — intravenous infusions 10 mg/kg on Day 1 of each 3-week cycle
  Other Names: cixutumumab; LY3012217
  Arms: Cohort 1, IMC A12 - 10 mg/kg
Biological: IMC-A12 (cixutumumab) - 20 mg/kg — intravenous infusions 20 mg/kg on Day 1 of each 3-week cycle
  Other Names: cixutumumab; LY3012217
  Arms: Cohort 2, IMC A12 20 - mg/kg
Drug: Sorafenib — 400 milligrams (mg) twice per day orally

SUMMARY:
To determine if IMC-A12 given in combination with Sorafenib is safe and effective for participants with advanced liver cancer.

DETAILED DESCRIPTION:
The purpose of this study is to determine progression-free survival (PFS) in participants with unresectable hepatocellular carcinoma who have received no prior systemic therapy when treated with IMC-A12 administered every three weeks in combination with oral sorafenib administered twice daily.

ELIGIBILITY:
Inclusion Criteria:

* The participant has histologically or cytologically confirmed, unresectable HCC
* The participant has at least one target lesion measurable according to Response Evaluation Criteria in Solid Tumors (RECIST) guidelines. Target lesion(s) must not lay within a previously irradiated, ablated, or chemoembolized area. If a lesion does lie in such an area, there must be evidence of growth on successive imaging studies, including tumor hypervascularity, in order for such a lesion to be considered a target lesion
* The participant has not received prior systemic therapy for HCC. Participants may have received prior embolization, chemoembolization, intra-arterial chemotherapy infusion, ethanol injection, radiofrequency ablation, or cryosurgery
* The participant has fasting serum glucose <160 milligrams/deciliter (mg/dL) or below the upper limit of normal (ULN) and/or hemoglobin A1C <7%. If baseline nonfasting glucose <160 mg/dL, fasting glucose measurement is not required
* The participant has the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* The participant has brain metastases
* The participant has acute hepatitis
* The participant has poorly controlled diabetes mellitus. Participants with a history of diabetes mellitus are allowed to participate, provided that their blood glucose is within normal range and that they are on a stable dietary or therapeutic regimen for this condition
* The participant has congestive heart failure > class II New York Heart Association (NYHA), unstable angina pectoris, new onset of angina pectoris, myocardial infarction within the past 6 months, or cardiac ventricular arrhythmias requiring antiarrhythmic therapy
* The participant has experienced a hemorrhage or bleeding event ≥ National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Grade 3 within 4 weeks prior first dose of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-05; Primary Completion 2012-10 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- United States (7):
  - ImClone Investigational Site, Scottsdale, Arizona
  - ImClone Investigational Site, Los Angeles, California
  - ImClone Investigational Site, Chicago, Illinois
  - ImClone Investigational Site, Metairie, Louisiana
  - ImClone Investigational Site, Burlington, Massachusetts
  - ImClone Investigational Site, New York, New York
  - ImClone Investigational Site, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who died or had progressive disease (PD) were considered to complete the study.
Groups:
- Cohort 1 - 10 mg/kg Cixutumumab: Cixutumumab (IMC-A12/LY3012217): 10 milligrams/kilogram (mg/kg) administered by intravenous (IV) infusion on Day 1 of each 3-week cycle.
  Sorafenib: 400 milligrams (mg) administered orally, twice daily on Days 1 through 21 of each 3-week cycle.
  Treatment cycles were repeated until there was evidence of PD, toxicity, or participant withdrawal.
- Cohort 2 - 20 mg/kg Cixutumumab: Cixutumumab: 20 mg/kg administered by IV infusions on Day 1 of each 3-week cycle
  Sorafenib: 400 mg administered orally, twice daily on Days 1 through 21 of each 3-week cycle
  Treatment cycles were repeated until there was evidence of PD, toxicity, or participant withdrawal.
Period: Overall Study
Arm/Group | Cohort 1 - 10 mg/kg Cixutumumab | Cohort 2 - 20 mg/kg Cixutumumab
Started | 6 | 41
Received Any Amount of Study Drug | 6 | 41
Completed | 6 | 33
Not Completed | 0 | 8
Not completed — Withdrawal by Subject | 0 | 5
Not completed — Other | 0 | 1
Not completed — Still on treatment at cutoff date | 0 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants who received any amount of study drug.
Groups:
- Cohort 1 - 10 mg/kg Cixutumumab: Cixutumumab: 10 mg/kg administered by IV infusion on Day 1 of each 3-week cycle.
  Sorafenib: 400 mg administered orally, twice daily on Days 1 through 21 of each 3-week cycle.
  Treatment cycles were repeated until there was evidence of PD, toxicity, or participant withdrawal.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - 10 mg/kg Cixutumumab | Cohort 2 - 20 mg/kg Cixutumumab | Total
Number analyzed (Participants) | 6 | 41 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (11.06) | 63.7 (8.79) | 64.2 (9.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 8 | 9
  Male | 5 | 33 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 8 | 9
  Not Hispanic or Latino | 5 | 33 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 7 | 7
  Black or African American | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 6 | 28 | 34
  Other | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 41 | 47

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from date of first dose of study drug until the date of objective PD or death due to any cause, whichever occurs first. PD defined as a ≥20% increase in the sum of the longest diameter (LD) of target lesions using as reference the smallest sum LD since baseline or ≥1 new lesions. Participants who died without PD were considered to have progressed on the date of death. Participants who were alive and without PD were censored at the time of the last objective tumor assessment. Participants who did not progress and are subsequently lost to follow-up were censored at the date of their last objective tumor assessment before loss to follow-up. Participants who progressed or died after ≥2 missed tumor assessment visits were censored at the date of their last objective tumor assessment before missed assessments. Participants who begin a new anticancer therapy were censored at the date of their last objective tumor assessment before initiation of new therapy.
Time Frame: Date of first dose of study drug up PD or death up to 12 months
Population: All randomized participants in Cohort 2 who received any amount of study drug, per the protocol efficacy analysis was only performed for Cohort 2. Participants censored = 10.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 2 - 20 mg/kg Cixutumumab
Number analyzed (Participants) | 41
months | 2.9 [1.7 to 5.3]

2. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Clinically significant events were defined as serious adverse events (SAEs) and other non-serious AEs regardless of causality. A summary of SAEs and other non-serious AEs regardless of causality, is located in the Reported Adverse Events module.
Time Frame: First day of treatment up to 22 months
Population: All randomized participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 10 mg/kg Cixutumumab | Cohort 2 - 20 mg/kg Cixutumumab
Number analyzed (Participants) | 6 | 41
Participants
  SAEs | 4 | 15
  Other Non-Serious AEs | 6 | 41

3. Secondary Outcome: Pharmacokinetic (PK): Maximum Concentration (Cmax) Cycle 1
Time Frame: Cycle 1, Day 1: Predose, 1 hour (h), 2 h, 168 h, 336 h, and 504 h after start of infusion (immediately prior to Cycle 2)
Population: Zero participants analyzed. No PK analysis was done, the assay used for PK assessment was not reliable and the values obtained could not be used. The samples expired before a new assay was developed, so data were not collected.
Arm/Group | Cohort 1 - 10 mg/kg Cixutumumab | Cohort 2 - 20 mg/kg Cixutumumab
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: PK: Minimum Concentration (Cmin) Cycle 1
Time Frame: Cycle 1, Day 1: Predose, 1 h, 2 h, 168 h, 336 h, and 504 h after start of infusion (immediately prior to Cycle 2)
Population: as for outcome 3
Arm/Group | Cohort 1 - 10 mg/kg Cixutumumab | Cohort 2 - 20 mg/kg Cixutumumab
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: PK: Half-Life (t1/2) Cycle 1
Time Frame: Cycle 1, Day 1: Predose, 1 h, 2 h, 168 h, 336 h, and 504 h after start of infusion (immediately prior to Cycle 2)
Population: as for outcome 3
Arm/Group | Cohort 1 - 10 mg/kg Cixutumumab | Cohort 2 - 20 mg/kg Cixutumumab
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: PK: Clearance (CL) Cycle 1
Time Frame: Cycle 1, Day 1: Predose, 1 h, 2 h, 168 h, 336 h, and 504 h after start of infusion (immediately prior to Cycle 2)
Population: as for outcome 3
Arm/Group | Cohort 1 - 10 mg/kg Cixutumumab | Cohort 2 - 20 mg/kg Cixutumumab
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: PK: Area Under the Concentration Versus Time Curve (AUC) Cycle 1
Time Frame: Cycle 1, Day 1: Predose, 1 h, 2 h, 168 h, 336 h, and 504 h after start of infusion (immediately prior to Cycle 2)
Population: as for outcome 3
Arm/Group | Cohort 1 - 10 mg/kg Cixutumumab | Cohort 2 - 20 mg/kg Cixutumumab
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: PK: Volume of Distribution at Steady State (Vss) Cycle 1
Time Frame: Cycle 1, Day 1: Predose, 1 h, 2 h, 168 h, 336 h, and 504 h after start of infusion (immediately prior to Cycle 2)
Population: as for outcome 3
Arm/Group | Cohort 1 - 10 mg/kg Cixutumumab | Cohort 2 - 20 mg/kg Cixutumumab
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: PK: Cmax Cycle 3
Time Frame: Cycle 3, Day 1: Predose, 2 h, 24 h, 48 h, 72 h, 168 h, 240 h, 336 h and 504 h after start of infusion (immediately prior to Cycle 4)
Population: as for outcome 3
Arm/Group | Cohort 1 - 10 mg/kg Cixutumumab | Cohort 2 - 20 mg/kg Cixutumumab
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: PK: Cmin Cycle 3
Time Frame: as for outcome 9
Population: as for outcome 3
Arm/Group | Cohort 1 - 10 mg/kg Cixutumumab | Cohort 2 - 20 mg/kg Cixutumumab
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: PK: t1/2 Cycle 3
Time Frame: as for outcome 9
Population: as for outcome 3
Arm/Group | Cohort 1 - 10 mg/kg Cixutumumab | Cohort 2 - 20 mg/kg Cixutumumab
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: PK: CL Cycle 3
Time Frame: as for outcome 9
Population: as for outcome 3
Arm/Group | Cohort 1 - 10 mg/kg Cixutumumab | Cohort 2 - 20 mg/kg Cixutumumab
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: PK: AUC Cycle 3
Time Frame: as for outcome 9
Population: as for outcome 3
Arm/Group | Cohort 1 - 10 mg/kg Cixutumumab | Cohort 2 - 20 mg/kg Cixutumumab
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: PK: Vss Cycle 3
Time Frame: as for outcome 9
Population: as for outcome 3
Arm/Group | Cohort 1 - 10 mg/kg Cixutumumab | Cohort 2 - 20 mg/kg Cixutumumab
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Percentage of Participants With Complete Response (CR) and Partial Response (PR) [Objective Response Rate (ORR)]
Description: Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST, version 1.0) criteria. CR was defined as the disappearance of all target and nontarget lesions and the normalization of tumor marker levels. PR was defined as having a ≥30% decrease in the sum of LD of target lesions taking as reference the baseline sum LD. Participants who did not have a tumor response assessment for any reason were considered nonresponders and were included in the denominator when calculating the response rate. Percentage of participants was calculated as: CR + PR / total number of participants in the treatment group * 100.
Time Frame: Date of first dose of study drug to PD up to 12 months
Population: All randomized participants in Cohort 2 who received any amount of study drug, per the protocol efficacy analysis was only performed for Cohort 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2 - 20 mg/kg Cixutumumab
Number analyzed (Participants) | 41
percentage of participants | 12.2 [4.1 to 26.2]

16. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of first dose of study drug to the date of death from any cause. If the participant was alive at the end of the follow-up period or was lost to follow-up, OS was censored on the last date the participant was known to be alive.
Time Frame: Date of first dose of study drug to date of death up to 22 months
Population: All randomized participants in Cohort 2 who received any amount of study drug, per the protocol efficacy analysis was only performed for Cohort 2. Participants censored = 19.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 2 - 20 mg/kg Cixutumumab
Number analyzed (Participants) | 41
months | 11.6 [8.0 to 15.1]

17. Secondary Outcome: Time to Disease Progression (TTP)
Description: TTP is defined as the time from the date of first dose of study drug until the date of objective disease progression. Participants without PD were censored at the time of the last objective tumor assessment. Participants who did not progress and lost to follow-up were censored at the date of the last objective tumor assessment before loss to follow-up. Participants who began new anticancer therapy prior to PD or death were censored at date of last tumor assessment prior to new therapy. Participants who died or had PD after ≥2 missed tumor assessments were censored at date of last tumor assessment prior to the missed assessments.
Time Frame: Date of first dose of study drug to date of PD up to 12 months
Population: All randomized participants in Cohort 2 who received any amount of study drug, per the protocol efficacy analysis was only performed for Cohort 2. Participants censored = 14.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 2 - 20 mg/kg Cixutumumab
Number analyzed (Participants) | 41
months | 3.0 [1.6 to 5.8]

18. Secondary Outcome: Duration of Response (DOR)
Description: Duration of CR or PR was defined as time from first objective assessment of CR or PR until first date of PD or death from any cause. Response was defined using RECIST v 1.0 criteria. CR was defined as disappearance of all target and nontarget lesions and normalization of tumor marker levels. PR was defined as a ≥30% decrease in the sum of LD of target lesions taking as reference the baseline sum LD. PD defined as a ≥20% increase in the sum of LD of target lesions using as reference the smallest sum LD since baseline or ≥1 new lesions. Participants with no PD, who discontinued treatment for toxicity or a reason other than PD, or were lost to follow-up, were censored at date of last tumor assessment. Participants who began new anticancer therapy prior to PD or death were censored at date of last tumor assessment prior to new therapy. Participants who died or had PD after ≥2 missed tumor assessments were censored at date of last tumor assessment prior to the missed assessments
Time Frame: Date of first occurrence of CR or PR to first date of PD or death up to 8 months
Population: All randomized participants in Cohort 2 who received any amount of study drug, per the protocol efficacy analysis was only performed for Cohort 2. Participants censored = 1.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 2 - 20 mg/kg Cixutumumab
Number analyzed (Participants) | 41
months | 7.1 [2.1 to 7.4]

19. Secondary Outcome: The Number of Participants With Serum Anti-Cixutumumab Antibody Assessment (Immunogenicity)
Description: A participant's serum sample was considered positive for antibodies against cixutumumab if it exhibited a post-treatment antibody level that exceeded the positive upper cut point determined from the anti-cixutumumab level seen in healthy untreated individuals. A participant was considered to have an anti-cixutumumab response if there were 2 consecutive positive samples or if the final sample tested was positive.
Time Frame: Predose, immediately prior to the first Cycle 3 and Cycle 5 infusions (3-week cycle) and 30 days after last dose of study drug
Population: Zero participants were analyzed. No assay was available to assess serum anti-cixutumumab antibodies.
Arm/Group | Cohort 1 - 10 mg/kg Cixutumumab | Cohort 2 - 20 mg/kg Cixutumumab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Cohort 1 - 10 mg/kg Cixutumumab: Cixutumumab: 10 mg/kg administered by IV infusion on Day 1 of each 3-week cycle.
  Sorafenib: 400 mg administered orally, twice per day on Days 1 through 21 of each 3-week cycle.
  Treatment cycles were repeated until there was evidence of PD, toxicity, or participant withdrawal.
- Cohort 2 - 20 mg/kg Cixutumumab: Cixutumumab: 20 mg/kg administered by IV infusions on Day 1 of each 3-week cycle.
  Sorafenib: 400 mg administered orally, twice per day on Days 1 through 21 of each 3-week cycle.
  Treatment cycles were repeated until there was evidence of PD, toxicity, or participant withdrawal.
Arm/Group | Cohort 1 - 10 mg/kg Cixutumumab | Cohort 2 - 20 mg/kg Cixutumumab
Serious Adverse Events (participants affected / at risk) | 4/6 | 15/41
Other Adverse Events (participants affected / at risk) | 6/6 | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - 10 mg/kg Cixutumumab (N=6) | Cohort 2 - 20 mg/kg Cixutumumab (N=41)
Retinal tear (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic haemorrhage (Hepatobiliary disorders) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cohort 1 - 10 mg/kg Cixutumumab (N=6) | Cohort 2 - 20 mg/kg Cixutumumab (N=41)
Anaemia (Blood and lymphatic system disorders) | 2 (4) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 4 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 12 (28)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 5 (5)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 8 (8)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 10 (12)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 18 (36)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 9 (9)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 10 (13)
Pancreatitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 2 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 10 (11)
Asthenia (General disorders) | 1 (1) | 2 (3)
Fatigue (General disorders) | 3 (9) | 25 (40)
Gait disturbance (General disorders) | 0 (0) | 3 (3)
Mucosal inflammation (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 4 (4)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (5) | 4 (5)
Candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 4 (4)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1/1 (1) | 0/8 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 5 (11)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 4 (11)
Blood albumin decreased (Investigations) | 1 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 3 (5)
Blood bilirubin increased (Investigations) | 0 (0) | 3 (3)
Blood creatinine increased (Investigations) | 2 (2) | 2 (2)
Lipase increased (Investigations) | 0 (0) | 8 (20)
Weight decreased (Investigations) | 1 (1) | 13 (14)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 16 (23)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 13 (26)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 9 (12)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 10 (15)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 7 (7)
Headache (Nervous system disorders) | 1 (2) | 7 (8)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3)
Confusional state (Psychiatric disorders) | 1 (2) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 5 (5)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Bladder pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 8 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 5 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 8 (8)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 15 (26)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 7 (12)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (5)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (2) | 4 (6)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 7 (8)

LIMITATIONS AND CAVEATS:
Per the protocol efficacy analysis was only performed for Cohort 2. No PK analysis was done, the assay used for PK assessment was not reliable and the values could not be used. The samples expired before a new assay was developed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.